CLINICAL TRIAL: NCT00148473
Title: A Single Dose of Oral Versus Vaginal Misoprostol for Induction of Labor: A Randomized Controlled Trial
Brief Title: Oral Versus Vaginal Misoprostol for Induction of Labor
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bangkok Metropolitan Administration Medical College and Vajira Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VJR-01
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2005-09-08 (Estimated); Status verified 2005-09

CONDITIONS: Termed Pregnancy With Indications for Labor Induction.
Keywords: Cervical ripening.; Induction of labor.; Misoprostol.
MeSH Terms: interventions — Misoprostol

INTERVENTIONS:
Drug: Misoprostol

SUMMARY:
The purpose of this study is to compare the efficacy between a single dose of oral misoprostol 100 microgram and vaginal misoprostol 50 microgram for induction of labor.

DETAILED DESCRIPTION:
Induction of labor is widely carried out all over the world in cases where continuation of pregnancy is hazardous to both the mother and/or fetus. The induction in a ripe cervix is not difficult but complications are significantly increased when the cervix is unripe. The only agent approved for cervical ripening and induction of labor in patients with an unripe cervix is dinoprostone(PGE2). Misoprostol is a synthetic PGE1 analogue marketed for the prevention and treatment of gastro-duodenal ulcers. Misoprostol costs much less than dinoprostone and does not require refrigeration and has few systemic side effects.In addition, it is rapidly absorbed orally and vaginally. Although misoprostol is not registered for such use, it has been widely used for obstetric indications such as induction of abortion and of labor. Misoprostol for induction of labor in preceding literatures mainly prescribed in multiple dosing regimen. The adverse effects on uterus potentially occur owing to the frequent administration of misoprostol. The objective of this study was to compare a single dose oral misoprostol with vaginal misoprostol.

ELIGIBILITY:
Inclusion Criteria:

* A live singleton pregnancy at a gestation of >37 weeks, with obstetric or medical indications for induction, and unfavorable cervix (the initial Bishop score of <717), vertex presentation, reactive fetal heart rate pattern, absence of labor, and intact membranes without previous stripping. Post-term inductions were considered when gestational age was >41 weeks.

Exclusion Criteria:

* Suspected cephalo-pelvic disproportion, estimated fetal weight of >4000 grams, maternal age of <18 years, parity of >5, previous cesarean delivery or history of uterine incision, any contraindication for vaginal delivery or prostaglandins administration and suspected chorioamnionitis.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180
Dates: Start 2000-03; Study Completion 2001-10

PRIMARY OUTCOMES:
The time interval from induction to vaginal delivery and vaginal delivery rate within 24 hours.

SECONDARY OUTCOMES:
Rate of vaginal delivery within 24 hours.
Cesarean section rate.
Uterine tachysystole.
Uterine hyperstimulation syndrome.
Number of women received oxytocin.
Neonatal outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Manit Sripramote, MD, Principal Investigator — BMA Medical College and Vajira Hospital
Locations (1):
- BMA Medical College and Vajira Hospital, Bangkok, Bangkok, Thailand